CLINICAL TRIAL: NCT01930916
Title: Accuracy of a Portable International Normalized Ratio Monitor in a Population Aged 75 Years Old and Over
Brief Title: Accuracy of a Portable International Normalized Ratio Monitor in Elderly Patients
Acronym: AGINR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-A00586-37
Record Dates: First submitted 2012-11-16; First posted 2013-08-29 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Blood Coagulation Disorders; Blood Coagulation Disorder With Prolonged Bleeding Time; Blood Coagulation Disorder With Prolonged Coagulation Time
Keywords: Prothrombin Time/instrumentation; Prothrombin Time/utilization; Blood Coagulation Disorders/blood; Blood Coagulation Disorders/complications; Blood Coagulation Disorders/diagnosis; Prospective Studies; Adult; Reproducibility of Results; Point-of-Care Systems/utilization; Aged; Elderly
MeSH Terms: conditions — Blood Coagulation Disorders; Disease; Patient Acceptance of Health Care | interventions — Antibodies, Antiphospholipid; Lupus Coagulation Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Not interventionnal (Other): INR capillary measurement with INRatio 2 device antiphospholipid antibodies and lupus anticoagulant
  Interventions: Device: INR capillary measurement with INRatio 2 device; Other: antiphospholipid antibodies and lupus anticoagulant

INTERVENTIONS:
Device: INR capillary measurement with INRatio 2 device — INR capillary measurement with INRatio 2 device
Other: antiphospholipid antibodies and lupus anticoagulant — Rate of antiphospholipid antibodies and lupus anticoagulant dosage A 5ml blood sample obtained by veinous punction.

SUMMARY:
Oral anticoagulants vitamin K antagonists (VKA) have been used for many years in the treatment of thromboembolic disorders, which are among the most costly diseases in terms of public health resources. According to the Agence française de sécurité sanitaire des produits de santé (AFSSAPS), it was estimated at about 900,000 the number of patients treated with VKA in 2008 (more than 1% of the French population). VKA are at the origin of many adverse effects, given their narrow therapeutic window. They are the cause of the death of approximately 5000 patients per year. The use of this therapy is a priority axis of reflection for the Haute Autorité de Santé.

The interregion G4 (Nord Pas de Calais, Normandy, Picardy), with more than 9 million people, is particularly affected by this problem.

University hospitals of our interregion, given their very substantial regional referral activity, are actually involved in managing VKA adverse side effects.

Elderly population constitutes the majority of prescriptions. The main objective of this study is to compare INR of people older than 75 years measured by traditional method with those measured by capillary method with INRatio2 supply.

The secondary objective is to show that this measure is not affected by the presence or absence of anti-phospholipid antibodies, probably very prevalent in the elderly, as well as to test the variability of INR measurement between different hospital.

DETAILED DESCRIPTION:
Adverse effects of oral anticoagulants (warfarin, fluindione mainly) are bleeding complications and concern 13% of hospitalizations, approximately 17,000 admissions per year. They constitute 12.3% of iatrogenic adverse effect according to the latest results of the survey conducted by the haute autorité de santé (HAS). A study realized in 2000, with 2976 patients, shows that 28.8% of patients were outside of any therapeutic range (<2 or> 4.5). In 2003, a third of french biologists had no knowledge of the indication of VKA treatment of patients at the INR measurement, and more than fifty percent in 2000. When the therapeutic range was known, the value of the INR remained outside it in 30% of cases. The median time between INR equilibration phase was 5 to 6 days, while the recommended time is 2 to 4 days. A quarter of patients in phase equilibrium treatment did not have a measure of INR at least once a month. Followed over a period of a year, patients spent 40% of the time with a value of INR outside the therapeutic range, high-risk area of recurrent thrombosis or hemorrhage. That is why they require regular monitoring of INR.

Currently, this monitoring is done through a blood sample analyzed by a laboratory according to standard techniques.

The use of the INR measurement by capillary method provides a result in less than 3 minutes. This also allows the development of different monitoring strategies. In the context of a self-monitoring measure, the patient himself performs the test using the device and therapeutic adjustment is made by the health care professional.

Data analysis by HAS showed that the use of a self-measurement device significantly improved the time spent in the therapeutic range, reduced the risk of major bleeding and the accident major thromboembolism.

The pathologies treated by VKA are more common in the elderly. They are also more vulnerable to falls, overdoses of these treatments because their pharmacokinetics is amended by polypharmacy, malnutrition, less protein binding. The relative risk of bleeding is multiplicated by two beyond 70 years. Despite the emergence of new anticoagulants in the prevention of complications of arrhythmia (this disorder affect nearly 10% of the population aged over 80 years), VKA remains prevalent because these new drugs have renal elimination that can not be monitored, and can not be dialysable, have no antidote and represent a daily cost about 30 times the VKA.

The question of the use of devices for self-measurement of INR in the elderly is particularly timely, because this population has never had, to our knowledge, a specific evaluation of this technique.

Elderly population would derive the greatest benefit of this system because it will significantly improve the time spend in the therapeutic range, and reduce the risk of bleeding and thromboembolic events in reducing INR fluctuations.

We build a multicenter study whose main objective is to demonstrate the concordance of INR measurement by the capillary way (INRatio2 ®, SAS ALERE, Jouy-en-Josas) with venous technical reference. It concerns patients older than 75 years treated with VKA and hospitalized in Internal Medicine, Geriatrics and Vascular Medicine in the fours university hospital of the G4 region. The secondary objectives are to estimate the prevalence of antiphospholipid antibodies (ranging from 12 to 55% depending on the study) and their influence on the measurement of the INR by capillary method and the variability of the INR veinous measurement in function of the hospital, with a centralized INR measurement which allow to compare. 150 patients is required to perform this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 75 years
* Recipient of the social security system
* Patient receiving anti vitamin K treatment
* Hospitalized in Internal Medicine, Geriatrics, Vascular Medicine
* Having signed an informed consent to participate in the study

Exclusion Criteria:

* Contraindication to a digital sampling.
* Conditions preventing the realization of INRatio2 ® test : Amputation of the extremities, trophic disorders of the extremities.
* Concomitant use of heparin.
* Mental or physical illness which do not permit to consent to participate in the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
INR by capillary method and INR by veinous punction | 24 hours
  INR by the classical way (punction) and comparison with a capillary method tested here.
  INR by capillary method is done immediately after inclusion. INR by veinous punction is done on the 24 hours after the inclusion.

SECONDARY OUTCOMES:
Difference between International normalized ratio (INR) measured in a veinous blood punction and with a capillary method on the same patient and correlated to the level of phospholipid antibodies and lupus anti coagulant | 1 year
  We want to know if the level of lupus and anti cardiolipin antibodies influence the value of INR measured by capillary method.
  lupus and anti cardiolipin antibodies tubes will be frozen after punction and analysed up to 1 year after.

OTHER OUTCOMES:
Difference of INR measurement by veinous method between Caen laboratory and the local center laboratory. | 1 year
  INR of a patient will be measured in two different center (Caen is the reference center).
  Blood sample will be frozen after punction and analysed up to 1 year after.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Bienvenu, M.D,Ph.D, Principal Investigator — Centre hospitalier régional universitaire de Caen; Jean Jacques Dutheil, Study Director — Centre hospitalier régional universitaire de Caen; Laurent Auboire, M.D, Study Chair — Centre hospitalier régional universitaire de Caen
Locations (4):
- France (4):
  - Centre hospitalier régional universitaire d'Amiens, Amiens
  - Centre hospitalier régional universitaire de Caen, Caen
  - Centre hospitalier régional universitaire de Lille, Lille
  - Centre hospitalier régional universitaire de Rouen, Rouen

REFERENCES:
- [Background] Manoussakis MN, Tzioufas AG, Silis MP, Pange PJ, Goudevenos J, Moutsopoulos HM. High prevalence of anti-cardiolipin and other autoantibodies in a healthy elderly population. Clin Exp Immunol. 1987 Sep;69(3):557-65. PMID 3499270
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. Population prevalence, incidence, and predictors of atrial fibrillation in the Renfrew/Paisley study. Heart. 2001 Nov;86(5):516-21. doi: 10.1136/heart.86.5.516. PMID 11602543
- [Background] Bazzan M, Montaruli B, Vaccarino A, Fornari G, Saitta M, Prandoni P. Presence of low titre of antiphospholipid antibodies in cancer patients: a prospective study. Intern Emerg Med. 2009 Dec;4(6):491-5. doi: 10.1007/s11739-009-0316-6. Epub 2009 Sep 26. PMID 19784751
- [Background] Sene D, Piette JC, Cacoub P. Antiphospholipid antibodies, antiphospholipid syndrome and infections. Autoimmun Rev. 2008 Feb;7(4):272-7. doi: 10.1016/j.autrev.2007.10.001. Epub 2007 Oct 23. PMID 18295729
- [Background] Quemeneur T, Lambert M, Hachulla E, Dubucquoi S, Caron C, Fauchais AL, Devulder B, Hatron PY. Significance of persistent antiphospholipid antibodies in the elderly. J Rheumatol. 2006 Aug;33(8):1559-62. PMID 16832847
- [Background] Perry SL, Samsa GP, Ortel TL. Point-of-care testing of the international normalized ratio in patients with antiphospholipid antibodies. Thromb Haemost. 2005 Dec;94(6):1196-202. doi: 10.1160/TH05-06-0400. PMID 16411394